CLINICAL TRIAL: NCT06078462
Title: Impact of Job Related Activities on Female Physiotherapist and Dentist During Internship Year
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Hend Reda Sakr, Lecturer of Physical Therapy for Woman's Health, Badr University
Other Study IDs: Hend4
Record Dates: First submitted 2022-11-16; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Job Related Stress
Keywords: hand grip; pinch grip; body composition; job related activities; physiotherapist; dentist
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Fifty physiotherapist females will participate in this group and will be assessed at the beginning of the study and after 6 months of clinical work.
  Interventions: Other: job related activities
- Group B: Fifty dentist females will participate in this group and will be assessed at the beginning of the study and after 6 months of clinical work.
  Interventions: Other: job related activities

INTERVENTIONS:
Other: job related activities — Different types of effort offered by female physiotherapist and female dentist during clinical practicing with patients in internship year

SUMMARY:
Response of hand grip, pinch grip and body composition to type of effort between female physiotherapist and female dentist at internship year.

DETAILED DESCRIPTION:
Fifty physiotherapist and fifty dentist females will be selected from faculty of physical therapy and faculty of dentistry at Badr University in Cairo BUC, both at internship year, and will be assigned into two groups. Group A consists of fifty physiotherapist females will participate in this group and will be assessed at the beginning of the study and after 6 months of clinical work. Group B consists of fifty dentist females will participate in this group and will be assessed at the beginning of the study and after 6 months of clinical work. Digital hand dynamometer will be used to assess hand grip strength and InBody device will be used to assess changes in body composition at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty physiotherapist females and fifty dentist females at internship year.
2. Their age will be ranged from 21 to 24 years old.
3. They are medically stable and consented to participate in the study.
4. They are able to follow instructions.

Exclusion Criteria:

1. History of any pathological disease-causing disorder in metabolism such as thyroid gland disorder.
2. History of muscular or neurological disorder.
3. Using any hormonal treatment.
4. Following any diet modification method.
5. Severe emotional stress.

Ages: 21 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifty physiotherapist and fifty dentist females will be selected from faculty of physical therapy and faculty of dentistry at Badr University in Cairo BUC
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Fist Grip | We measure fist grip at 1st time at the beginning of work as interns in clinic then we re-measure fist grip again to assess its progression after 6 months of work..
  Maximum grip value using hand held dynamometer
Lateral Pinch (key pinch) | We measure lateral pinch at 1st time at the beginning of work as interns in clinic then we re-measure lateral pinch again to assess its progression after 6 months of work.
  using Jamar pinch guage
Palmer pinch (chunk pinch) | We measure lateral pinch at 1st time at the beginning of work as interns in clinic then we re-measure lateral pinch again to assess its progression after 6 months of work..
  using Jamar pinch guage
Pulp to pulp | We measure pulp to pulp grip at 1st time at the beginning of work as interns in clinic then we re-measure pulp to pulp grip again to assess its progression after 6 months of work..
  using Jamar pinch guage
Tip to tip | We measure tip to tip grip at 1st time at the beginning of work as interns in clinic then we re-measure tip to tip grip again to assess its progression after 6 months of work..
  using Jamar pinch guage
Body mass index | We measure obesity index at 1st time at the beginning of work as interns in clinic then we re-measure obesity index again to assess its progression after 6 months of work..
  Using INBODY device
Percent of body fat in kg | We measure percent of body fat at 1st time at the beginning of work as interns in clinic then we re-measure percent of body fat again to assess its progression after 6 months of work..
  Using INBODY device
Lean muscle mass in kg | We measure percent of muscle mass at 1st time at the beginning of work as interns in clinic then we re-measure percent of muscle mass again to assess its progression after 6 months of work..
  Using INBODY device

CONTACTS AND LOCATIONS:
Overall Officials: Hend R Sakr, Principal Investigator — Lecturer of Physical Therapy for Women's Health, Badr University in Cairo BUC
Locations (2):
- Egypt (2):
  - Badr University in Cairo, New Cairo, Badr City
  - Faculty of Physical Therapy, Badr University, Cairo, New Cairo

IPD SHARING:
Plan to Share IPD: Undecided